CLINICAL TRIAL: NCT01368250
Title: SwissTAVI Registry: Prospective, National, Multi-Center Registry of Patients Undergoing Transcatheter Aortic Valve Implantation
Brief Title: SwissTAVI Registry
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 056/11
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Aortic Valve Disease Mixed
Keywords: Aortic valve; Heart valve; VARC; Transcatheter; Minimal-invasive; TAVI; TAVR
MeSH Terms: interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Patients with native aortic stenosis undergoing TAVI
  Interventions: Procedure: Transcatheter Aortic Valve Implantation
- 2: Patients with native aortic regurgitation undergoing TAVI
- 3: Patients with degenerative surgical bioprosthesis undergoing TAV-in-SAV

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Implantation — Minimal Invasive Implantation of a biological prosthesis in Aortic Position
  Groups: 1

SUMMARY:
The purpose of this prospective multi-center, observational national registry in Switzerland is to obtain clinical baseline, procedural and follow-up data of all patients treated with TAVI in Switzerland and to assess short, mid- and long-term clinical outcome data of the CE approved devices. All centers in Switzerland implanting the CE approved devices for TAVI will be invited to include patients in the registry. Each site will collect baseline and procedural data as well as clinical outcome data up to five years.

DETAILED DESCRIPTION:
The present registry aims to assess the safety and efficacy of TAVI with CE approved devices at Swiss cardiovascular centers. The Swiss Working group of Interventional Cardiology and Acute Coronary Syndrome decided to establish a nationwide registry in collaboration with the Swiss Society of Cardiac Surgery in order to assess the procedural and clinical outcome of TAVI patients. This prospective registry will help to identify candidates for TAVI, will report on peri-procedural outcome and on long-term efficacy of the devices. Last but not least it is a tool to increase quality of treatment of this high-risk patient population.

Methods

This is a prospective multi-center, observational registry performed in Switzerland. All centers in Switzerland implanting the CE approved devices for TAVI will be invited to consecutively include patients in the registry. Each center will sign an agreement that all patients will be included in the registry. Each site will collect baseline and procedural data as well as clinical outcome data up to 15 years after TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Native aortic valve stenosis
* Native aortic valve regurgitation
* Degenerated aortic bioprosthesis requiring treatment

Exclusion Criteria

* Patients refuses informed consent to participate in the registry
* Contraindication for TAVI
* High probability of non-adherence to the follow up - requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with aortic valve disease or degenerated aortic bioprosthesis scheduled to undergo transcatheter aortic valve implantation (TAVI) using commercially available devices with CE approval are eligible for enrollment in the registry. The TAVI procedure can be performed using all available access routes.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2011-02; Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
combined early safety and clinical efficacy as defined by the Valve Academic Research Consortium-2 (VARC-2) | 1 year
  Composed by:
  * death
  * stroke
  * aortic valve re-intervention
  * structural valve deterioration
  * myocardial Infarction

SECONDARY OUTCOMES:
combined early safety and clinical efficacy as defined by the Valve Academic Research Consortium-2 (VARC-2) | 30days
  Composed by:
  * death
  * stroke
  * aortic valve re-intervention
  * myocardial Infarction
  * kidney injury
  * access related complications
  * pacemaker requirements
combined safety and clinical efficacy as defined by the Valve Academic Research Consortium-2 (VARC-2) | 5 years
  Composed by:
  * death
  * stroke
  * aortic valve re-intervention
  * structural valve deterioration
combined safety and clinical efficacy as defined by the Valve Academic Research Consortium-2 (VARC-2) | 10 years , 15 years
  Composed by:
  * death
  * stroke
  * aortic valve re-intervention
  * structural valve deterioration

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Stortecky, MD, Study Chair — Bern University Hospital
Locations (1):
- Department of Cardiology, Bern, Switzerland

REFERENCES:
- [Derived] Tomii D, Alaour B, Heg D, Okuno T, Nakase M, Samim D, Praz F, Lanz J, Stortecky S, Reineke D, Windecker S, Pilgrim T. Self-expanding versus balloon-expandable transcatheter heart valves in patients with excessive aortic valve cusp calcification. Am Heart J. 2026 Feb;292:107279. doi: 10.1016/j.ahj.2025.09.011. Epub 2025 Sep 18. PMID 40975195
- [Derived] Badertscher P, Stortecky S, Serban T, Knecht S, Heg D, Tueller D, Jeger R, Reuthebuch O, Muller O, Toggweiler S, Wenaweser P, Huber C, Roffi M, Ferrari E, Reichlin T, Nestelberger T, Mahfoud F, Kuhne M, Sticherling C; SwissTAVI Investigators. Long-Term Outcomes of Patients Requiring Pacemaker Implantation After Transcatheter Aortic Valve Replacement: The SwissTAVI Registry. JACC Cardiovasc Interv. 2025 May 12;18(9):1163-1171. doi: 10.1016/j.jcin.2025.03.028. Epub 2025 Apr 1. PMID 40368460
- [Derived] Nakase M, Draxler DF, Tomii D, Heg D, Okuno T, Samim D, Lanz J, Stortecky S, Reineke D, Windecker S, Pilgrim T. Incidence, predictors and clinical impact of upper gastrointestinal bleeding after transcatheter aortic valve replacement. Heart. 2025 Nov 12;111(23):1149-1155. doi: 10.1136/heartjnl-2024-325359. PMID 40348411
- [Derived] Tomii D, Heg D, Nakase M, Samim D, Lanz J, Praz F, Stortecky S, Reineke D, Windecker S, Pilgrim T. Flow Status-Based Predicted Prosthesis-Patient Mismatch in Patients Undergoing Transcatheter Aortic Valve Replacement With a Balloon-Expandable Valve. Struct Heart. 2024 Dec 6;9(4):100379. doi: 10.1016/j.shj.2024.100379. eCollection 2025 Apr. PMID 40321306
- [Derived] Nakase M, Tomii D, Maznyczka A, Heg D, Okuno T, Samim D, Stortecky S, Lanz J, Reineke D, Windecker S, Pilgrim T. Five-year outcomes with self-expanding versus balloon-expandable TAVI in patients with left ventricular systolic dysfunction. Am Heart J. 2025 Feb;280:18-29. doi: 10.1016/j.ahj.2024.10.018. Epub 2024 Nov 12. PMID 39536846
- [Derived] Nakase M, Tomii D, Samim D, Grani C, Praz F, Lanz J, Stortecky S, Reineke D, Windecker S, Pilgrim T. Impact of Severity and Extent of Iliofemoral Atherosclerosis on Clinical Outcomes in Patients Undergoing TAVR. JACC Cardiovasc Interv. 2024 Oct 28;17(20):2353-2363. doi: 10.1016/j.jcin.2024.07.009. Epub 2024 Oct 9. PMID 39387783
- [Derived] Tomii D, Heg D, Lanz J, Nakase M, Samim D, Stortecky S, Reineke D, Windecker S, Pilgrim T. Renin-Angiotensin System Inhibition in Patients With Myocardial Injury Complicating Transcatheter Aortic Valve Replacement. JACC Adv. 2024 Aug 16;3(9):101212. doi: 10.1016/j.jacadv.2024.101212. eCollection 2024 Sep. PMID 39253713
- [Derived] Tomii D, Okuno T, Nakase M, Praz F, Stortecky S, Reineke D, Windecker S, Lanz J, Pilgrim T. Renin-Angiotensin System Inhibition and Cardiac Damage in Patients Undergoing Transcatheter Aortic Valve Replacement. Can J Cardiol. 2024 Dec;40(12):2592-2602. doi: 10.1016/j.cjca.2024.07.019. Epub 2024 Jul 25. PMID 39067618
- [Derived] Nakase M, Tomii D, Maznyczka A, Samim D, Lanz J, Praz F, Stortecky S, Reineke D, Windecker S, Pilgrim T. Sex-Specific Differences in Upstream Cardiac Damage in Patients With Aortic Stenosis Undergoing TAVR. JACC Cardiovasc Interv. 2024 May 27;17(10):1252-1264. doi: 10.1016/j.jcin.2024.03.031. PMID 38811107
- [Derived] Nakase M, Tomii D, Heg D, Praz F, Stortecky S, Reineke D, Samim D, Lanz J, Windecker S, Pilgrim T. Long-Term Impact of Cardiac Damage Following Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2024 Apr 22;17(8):992-1003. doi: 10.1016/j.jcin.2024.02.011. PMID 38658128
- [Derived] Alaour B, Ferrari E, Heg D, Tueller D, Pilgrim T, Muller O, Noble S, Jeger R, Reuthebuch O, Toggweiler S, Templin C, Wenaweser P, Nietlispach F, Taramasso M, Huber C, Roffi M, Windecker S, Stortecky S. Non-Vitamin K Antagonist Versus Vitamin K Antagonist Oral Anticoagulant Agents After Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2024 Feb 12;17(3):405-418. doi: 10.1016/j.jcin.2023.11.038. PMID 38355269
- [Derived] Okuno T, Alaour B, Heg D, Tueller D, Pilgrim T, Muller O, Noble S, Jeger R, Reuthebuch O, Toggweiler S, Ferrari E, Templin C, Wenaweser P, Nietlispach F, Taramasso M, Huber C, Roffi M, Windecker S, Stortecky S. Long-Term Risk of Stroke After Transcatheter Aortic Valve Replacement: Insights From the SwissTAVI Registry. JACC Cardiovasc Interv. 2023 Dec 25;16(24):2986-2996. doi: 10.1016/j.jcin.2023.10.021. PMID 38151313
- [Derived] Tomii D, Okuno T, Heg D, Nakase M, Lanz J, Praz F, Stortecky S, Reineke D, Windecker S, Pilgrim T. Long-term outcomes of measured and predicted prosthesis-patient mismatch following transcatheter aortic valve replacement. EuroIntervention. 2023 Nov 17;19(9):746-756. doi: 10.4244/EIJ-D-23-00456. PMID 37622754
- [Derived] Nakase M, Tomii D, Heg D, Praz F, Stortecky S, Lanz J, Reineke D, Windecker S, Pilgrim T. Association of atrial fibrillation with survival in patients with low-flow low-gradient aortic stenosis with preserved ejection fraction undergoing TAVI. Eur Heart J Qual Care Clin Outcomes. 2024 May 22;10(3):246-255. doi: 10.1093/ehjqcco/qcad045. PMID 37491693
- [Derived] Alwan L, Tomii D, Heg D, Okuno T, Lanz J, Praz F, Chong-Nguyen C, Stortecky S, Reineke D, Windecker S, Pilgrim T. Impact of right ventricular-pulmonary arterial coupling on clinical outcomes in patients undergoing transcatheter aortic valve implantation. Cardiovasc Revasc Med. 2023 Nov;56:27-34. doi: 10.1016/j.carrev.2023.05.008. Epub 2023 May 16. PMID 37210220
- [Derived] Okuno T, Tomii D, Lanz J, Heg D, Praz F, Stortecky S, Reineke D, Windecker S, Pilgrim T. 5-Year Outcomes With Self-Expanding vs Balloon-Expandable Transcatheter Aortic Valve Replacement in Patients With Small Annuli. JACC Cardiovasc Interv. 2023 Feb 27;16(4):429-440. doi: 10.1016/j.jcin.2022.11.032. PMID 36858662
- [Derived] Tomii D, Okuno T, Lanz J, Stortecky S, Reineke D, Windecker S, Pilgrim T. Valve-in-valve TAVI and risk of coronary obstruction: Validation of the VIVID classification. J Cardiovasc Comput Tomogr. 2023 Mar-Apr;17(2):105-111. doi: 10.1016/j.jcct.2023.01.042. Epub 2023 Feb 6. PMID 36754691
- [Derived] Tomii D, Okuno T, Lanz J, Stortecky S, Windecker S, Pilgrim T. Aortic annulus ellipticity and outcomes after transcatheter aortic valve implantation. Catheter Cardiovasc Interv. 2023 Jan;101(1):199-208. doi: 10.1002/ccd.30507. Epub 2022 Dec 1. PMID 36453455
- [Derived] Okuno T, Demirel C, Tomii D, Heg D, Haner J, Siontis GCM, Lanz J, Raber L, Strotecky S, Furholz M, Praz F, Windecker S, Pilgrim T. Long-term risk of unplanned percutaneous coronary intervention after transcatheter aortic valve replacement. EuroIntervention. 2022 Nov 18;18(10):797-803. doi: 10.4244/EIJ-D-22-00342. PMID 36039573
- [Derived] Mergen V, Sartoretti T, Baer-Beck M, Schmidt B, Petersilka M, Wildberger JE, Euler A, Eberhard M, Alkadhi H. Ultra-High-Resolution Coronary CT Angiography With Photon-Counting Detector CT: Feasibility and Image Characterization. Invest Radiol. 2022 Dec 1;57(12):780-788. doi: 10.1097/RLI.0000000000000897. Epub 2022 May 31. PMID 35640019
- [Derived] Okuno T, Tomii D, Buffle E, Lanz J, Ryffel C, Demirel C, Hashemi S, Hagemeyer D, Papadis A, Heg D, Praz F, Stortecky S, Windecker S, Pilgrim T. Transcatheter aortic valve implantation in patients with rheumatic aortic stenosis. Heart. 2022 Jul 13;108(15):1225-1233. doi: 10.1136/heartjnl-2021-320531. PMID 35351823
- [Derived] Tomii D, Okuno T, Demirel C, Praz F, Lanz J, Stortecky S, Windecker S, Pilgrim T. Impact of First-Phase Ejection Fraction on Clinical Outcomes in Patients Undergoing Transcatheter Aortic Valve Implantation. Cardiovasc Revasc Med. 2022 Sep;42:55-61. doi: 10.1016/j.carrev.2022.02.023. Epub 2022 Feb 26. PMID 35283064
- [Derived] Tomii D, Okuno T, Heg D, Lanz J, Praz F, Stortecky S, Windecker S, Pilgrim T. Validation of the VARC-3 Technical Success Definition in Patients Undergoing TAVR. JACC Cardiovasc Interv. 2022 Feb 28;15(4):353-364. doi: 10.1016/j.jcin.2021.11.013. Epub 2022 Jan 31. PMID 35093281
- [Derived] Mergen V, Sartoretti T, Klotz E, Schmidt B, Jungblut L, Higashigaito K, Manka R, Euler A, Kasel M, Eberhard M, Alkadhi H. Extracellular Volume Quantification With Cardiac Late Enhancement Scanning Using Dual-Source Photon-Counting Detector CT. Invest Radiol. 2022 Jun 1;57(6):406-411. doi: 10.1097/RLI.0000000000000851. Epub 2022 Jan 21. PMID 35066531
- [Derived] Okuno T, Tomii D, Heg D, Lanz J, Praz F, Stortecky S, Reineke D, Windecker S, Pilgrim T. Five-year outcomes of mild paravalvular regurgitation after transcatheter aortic valve implantation. EuroIntervention. 2022 May 15;18(1):33-42. doi: 10.4244/EIJ-D-21-00784. PMID 34930717
- [Derived] Tomii D, Okuno T, Heg D, Grani C, Lanz J, Praz F, Stortecky S, Windecker S, Pilgrim T, Reineke D. Sinus of Valsalva Dimension and Clinical Outcomes in Patients Undergoing Transcatheter Aortic Valve Implantation. Am Heart J. 2022 Feb;244:94-106. doi: 10.1016/j.ahj.2021.11.004. Epub 2021 Nov 14. PMID 34788603
- [Derived] Tomii D, Okuno T, Praz F, Heg D, Wild MG, Lanz J, Stortecky S, Reineke D, Windecker S, Pilgrim T. Potential Candidates for Transcatheter Tricuspid Valve Intervention After Transcatheter Aortic Valve Replacement: Predictors and Prognosis. JACC Cardiovasc Interv. 2021 Oct 25;14(20):2246-2256. doi: 10.1016/j.jcin.2021.07.030. Epub 2021 Sep 29. PMID 34600873
- [Derived] Okuno T, Lanz J, Stortecky S, Heg D, Bernhard B, Grani C, Huber A, Praz F, Raber L, Valgimigli M, Siontis GCM, Windecker S, Pilgrim T. Clinical impact of left atrial appendage filling defects in patients undergoing transcatheter aortic valve implantation. Eur Heart J Cardiovasc Imaging. 2022 Sep 10;23(10):1354-1364. doi: 10.1093/ehjci/jeab142. PMID 34463717
- [Derived] Eberhard M, Hinzpeter R, Schonenberger ALN, Euler A, Kuzo N, Reeve K, Stahli BE, Kasel AM, Manka R, Tanner FC, Alkadhi H. Incremental Prognostic Value of Coronary Artery Calcium Score for Predicting All-Cause Mortality after Transcatheter Aortic Valve Replacement. Radiology. 2021 Oct;301(1):105-112. doi: 10.1148/radiol.2021204623. Epub 2021 Aug 3. PMID 34342499
- [Derived] Okuno T, Heg D, Lanz J, Praz F, Brugger N, Stortecky S, Windecker S, Pilgrim T. Refined staging classification of cardiac damage associated with aortic stenosis and outcomes after transcatheter aortic valve implantation. Eur Heart J Qual Care Clin Outcomes. 2021 Oct 28;7(6):532-541. doi: 10.1093/ehjqcco/qcab041. PMID 34086888
- [Derived] Attinger-Toller A, Ferrari E, Tueller D, Templin C, Muller O, Nietlispach F, Toggweiler S, Noble S, Roffi M, Jeger R, Huber C, Carrel T, Pilgrim T, Wenaweser P, Togni M, Cook S, Heg D, Windecker S, Goy JJ, Stortecky S. Age-Related Outcomes After Transcatheter Aortic Valve Replacement: Insights From the SwissTAVI Registry. JACC Cardiovasc Interv. 2021 May 10;14(9):952-960. doi: 10.1016/j.jcin.2021.01.042. Epub 2021 Apr 14. PMID 33865734
- [Derived] Okuno T, Corpataux N, Spano G, Grani C, Heg D, Brugger N, Lanz J, Praz F, Stortecky S, Siontis GCM, Windecker S, Pilgrim T. True-severe stenosis in paradoxical low-flow low-gradient aortic stenosis: outcomes after transcatheter aortic valve replacement. Eur Heart J Qual Care Clin Outcomes. 2021 Jul 21;7(4):366-377. doi: 10.1093/ehjqcco/qcab010. PMID 33576388
- [Derived] Sweda R, Dobner S, Heg D, Lanz J, Malebranche D, Langhammer B, Okuno T, Praz F, Raber L, Valgimigli M, Reineke D, Pilgrim T, Windecker S, Stortecky S. Discharge Location and Outcomes After Transcatheter Aortic Valve Implantation. Am J Cardiol. 2021 Feb 1;140:95-102. doi: 10.1016/j.amjcard.2020.10.058. Epub 2020 Nov 2. PMID 33144166
- [Derived] Okuno T, Brugger N, Asami M, Heg D, Siontis GCM, Winkel MG, Lanz J, Grani C, Huber A, Stortecky S, George I, Kodali S, Pilgrim T, Windecker S, Khalique OK, Praz F. Clinical impact of mitral calcium volume in patients undergoing transcatheter aortic valve implantation. J Cardiovasc Comput Tomogr. 2021 Jul-Aug;15(4):356-365. doi: 10.1016/j.jcct.2020.10.003. Epub 2020 Oct 21. PMID 33121904
- [Derived] Okuno T, Hagemeyer D, Brugger N, Ryffel C, Heg D, Lanz J, Praz F, Stortecky S, Raber L, Roten L, Reichlin T, Windecker S, Pilgrim T. Valvular and Nonvalvular Atrial Fibrillation in Patients Undergoing Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2020 Sep 28;13(18):2124-2133. doi: 10.1016/j.jcin.2020.05.049. PMID 32972574
- [Derived] Okuno T, Asami M, Heg D, Lanz J, Praz F, Hagemeyer D, Brugger N, Grani C, Huber A, Spirito A, Raber L, Stortecky S, Windecker S, Pilgrim T. Impact of Left Ventricular Outflow Tract Calcification on Procedural Outcomes After Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2020 Aug 10;13(15):1789-1799. doi: 10.1016/j.jcin.2020.04.015. PMID 32763071
- [Derived] Stortecky S, Heg D, Tueller D, Pilgrim T, Muller O, Noble S, Jeger R, Toggweiler S, Ferrari E, Taramasso M, Maisano F, Hoeller R, Wenaweser P, Nietlispach F, Widmer A, Huber C, Roffi M, Carrel T, Windecker S, Conen A. Infective Endocarditis After Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2020 Jun 23;75(24):3020-3030. doi: 10.1016/j.jacc.2020.04.044. PMID 32553254
- [Derived] Muller O, Fournier S, Pilgrim T, Heg D, Noble S, Jeger R, Toggweiler S, Taramasso M, Windecker S, Stortecky S; SwissTAVI Investigators. Local Versus General Anesthesia for Transcatheter Aortic Valve Replacement: A SwissTAVI Registry Analysis. JACC Cardiovasc Interv. 2019 Sep 23;12(18):1874-1876. doi: 10.1016/j.jcin.2019.05.047. No abstract available. PMID 31537296
- [Derived] Baumann F, Obeid S, Gilhofer T, Siegrist P, von Spiczak J, Luscher TF, Binder RK. Right coronary artery motion analysis: a novel method to measure right ventricular systolic function by selective coronary angiography. Int J Cardiovasc Imaging. 2019 Sep;35(9):1557-1561. doi: 10.1007/s10554-019-01606-9. Epub 2019 May 2. PMID 31044328
- [Derived] Asami M, Pilgrim T, Lanz J, Heg D, Franzone A, Piccolo R, Langhammer B, Praz F, Raber L, Valgimigli M, Roost E, Windecker S, Stortecky S. Prognostic Relevance of Left Ventricular Myocardial Performance After Transcatheter Aortic Valve Replacement. Circ Cardiovasc Interv. 2019 Jan;12(1):e006612. doi: 10.1161/CIRCINTERVENTIONS.118.006612. PMID 30626203
- [Derived] Asami M, Stortecky S, Praz F, Lanz J, Raber L, Franzone A, Piccolo R, Siontis GCM, Heg D, Valgimigli M, Wenaweser P, Roost E, Windecker S, Pilgrim T. Prognostic Value of Right Ventricular Dysfunction on Clinical Outcomes After Transcatheter Aortic Valve Replacement. JACC Cardiovasc Imaging. 2019 Apr;12(4):577-587. doi: 10.1016/j.jcmg.2017.12.015. Epub 2018 Feb 14. PMID 29454762
- [Derived] Binder RK, Stortecky S, Heg D, Tueller D, Jeger R, Toggweiler S, Pedrazzini G, Amann FW, Ferrari E, Noble S, Nietlispach F, Maisano F, Raber L, Roffi M, Grunenfelder J, Juni P, Huber C, Windecker S, Wenaweser P. Procedural Results and Clinical Outcomes of Transcatheter Aortic Valve Implantation in Switzerland: An Observational Cohort Study of Sapien 3 Versus Sapien XT Transcatheter Heart Valves. Circ Cardiovasc Interv. 2015 Oct;8(10):e002653. doi: 10.1161/CIRCINTERVENTIONS.115.002653. PMID 26453687
- [Derived] Wenaweser P, Stortecky S, Heg D, Tueller D, Nietlispach F, Falk V, Pedrazzini G, Jeger R, Reuthebuch O, Carrel T, Raber L, Amann FW, Ferrari E, Toggweiler S, Noble S, Roffi M, Gruenenfelder J, Juni P, Windecker S, Huber C. Short-term clinical outcomes among patients undergoing transcatheter aortic valve implantation in Switzerland: the Swiss TAVI registry. EuroIntervention. 2014 Dec;10(8):982-9. doi: 10.4244/EIJV10I8A166. PMID 24694729